CLINICAL TRIAL: NCT04027595
Title: Neodymium-doped Yttrium Aluminum Garnet (Nd: YAG) Laser Capsulotomy: Efficacy and Outcomes Performed by Optometrists
Brief Title: Efficacy and Outcomes of Neodymium-doped Yttrium Aluminum Garnet (Nd: YAG) Laser Capsulotomy Performed by Optometrists
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Northeastern State University (Other)
Responsible Party: Sponsor
Other Study IDs: NSUOCO2020
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Posterior Capsule Opacification Obscuring Vision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Neodymium-doped Yttrium Aluminum Garnet (Nd: YAG) Laser Capsulotomy — A Nd: YAG laser will be used to open the cloudy posterior capsule of the lens to improve central visual acuity.

SUMMARY:
The purpose of this study is to formally assess the efficacy and outcomes of optometrist-performed neodymium-doped yttrium aluminum garnet (Nd: YAG) laser capsulotomy procedures.

DETAILED DESCRIPTION:
Participants will undergo a pre-procedure examination to establish baseline findings and to determine if they meet the inclusion criteria. Participants will undergo the Nd: YAG laser capsulotomy procedure and will be examined at 1 hour, 1 day (if necessary), 1 week, 1 month, and 3 months following the procedure. Follow-up examinations will evaluate visual acuity improvement and possible post-procedure complications. The complication rate following the laser capsulotomy procedure is typically minimal.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent;
2. At least 18 years of age, male or female;
3. Prior cataract surgery;
4. Diagnosed with posterior capsule opacification obstructing vision;
5. Best-corrected visual acuity less than 20/40 or visual acuity with glare that reduces by 2 lines or more on an ETDRS visual acuity chart or significant effect on activities of daily living

Exclusion Criteria:

1. History of underlying ocular disease (not including mild/moderate non-proliferative diabetic retinopathy or incidental findings)
2. Previous myopic refractive error greater than 6.00 diopters
3. Complications following previous ocular procedures (i.e. intraocular lens decentration)
4. Ocular surgery other than uncomplicated cataract or uncomplicated refractive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Existing patients at primary eye care optometric facilities.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Central Visual Acuity | 3 months
  Pre and Post Procedure Visual Acuity

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Lighthizer, OD, Study Director — Northeastern State University
Locations (1):
- Northeastern State University, Tahlequah, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided